CLINICAL TRIAL: NCT05428761
Title: A Randomized, Placebo Controlled, Semi-Blind, Crossover Study to Evaluate the Effects of Two Novel Hydration Beverage Formulas on Rehydration in Healthy Adults
Brief Title: Clinical Trial to Evaluate the Effects of Two Novel Hydration Beverage Formulas on Rehydration in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liquid I.V. (Other)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network); University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: SOW4
Record Dates: First submitted 2022-06-15; First posted 2022-06-23 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Dehydration; Rehydration; Exercise Performance; Exercise Recovery; Fluid Balance; Cognitive Performance
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TP1 (Experimental): Participants will receive TP1 during one experimental trial.
  Interventions: Other: TP1
- TP2 (Experimental): Participants will receive TP2 during one experimental trial.
  Interventions: Other: TP2
- Placebo (Placebo Comparator): Participants will receive placebo during one experimental trial.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: TP1 — Participants will receive TP1 during one experimental visit.
  Arms: TP1
Other: TP2 — Participants will receive TP2 during one experimental visit.
  Arms: TP2
Other: Placebo — Participants will receive placebo during one experimental visit.
  Arms: Placebo

SUMMARY:
Dehydration lowers both physical and mental performance if it is severe enough. Performance declines are more pronounced in hot conditions or after prolonged strenuous activity such as exercise. Most individuals drink less than their sweat losses during activity, while some individuals overdrink and develop a sodium deficiency.

Water and electrolyte balance must be restored as part of the recovery process after any activity that causes sweating. Plain water causes a decrease in plasma sodium concentration and osmolality, which reduces the desire to drink and increases urine production. Unless the volume ingested exceeds the loss, individuals are in net negative fluid balance throughout the recovery period due to urinary losses. When sodium and potassium are added to rehydration fluids, urine production is reduced in the hours following rehydration. Rehydration is only possible if a volume of fluid equal to or greater than the amount lost through sweat is consumed, together with adequate electrolytes.

The test products for this study, TP1 and TP2, are novel hydration beverage formulas. They are an electrolyte drink mixture with five essential vitamins and three times more electrolytes than typical sports beverages. The test products create an osmotic force that permits water to be supplied to the bloodstream sooner in the digestive system by using a specific ratio of sodium, glucose, and potassium. This randomized, placebo-controlled, semi-blind, crossover study will evaluate the effects of the test products on rehydration in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female participants who are between 18 and 49 years of age (inclusive).
* Are in good general health (no active or uncontrolled diseases or conditions) and can ingest the assigned amount of fluid at each visit.
* Have a body mass index (BMI) between 17.0 and 29.9 kg/m2 (inclusive).
* Exercise regularly as per physical activity guidelines for Americans [structured exercise for a minimum of 150 cumulative minutes per week (low end) to 500 cumulative minutes of exercise per week (high-end)] and willing to maintain the same level of physical activity throughout the study period.
* Can maintain their exercise status at the beginning of the study throughout the study period.
* Can achieve a peak VO2 at screening that is at least 60% of their age and gender matched normative value per American College of Sports Medicine recommendations.
* Have normal or acceptable to to the investigator vital signs (BP and HR) at screening.
* Individuals with childbearing potential:
* Agree to practice an acceptable form of birth control for a certain timeframe prior to the first dose of study product and throughout the study, including:

  1. use for at least three months prior to the first dose of study product: hormonal contraceptives including oral contraceptives, hormone birth control patch (e.g., Ortho Evra), vaginal contraceptive ring (e.g., NuvaRing), injectable contraceptives (e.g., Depo-Provera, Lunelle), hormonal intrauterine devices (e.g., Mirena), or hormone implant (e.g., Norplant System); or
  2. use for at least one month prior to the first dose of study product: double-barrier method, non-hormonal intrauterine devices (i.e., copper), or complete abstinence from sexual intercourse that can result in pregnancy; or
  3. vasectomy of partner at least six months prior to the first dose of study product.
* Individuals with the potential to impregnate others:
* Agree to use condom or other acceptable methods to prevent pregnancy throughout the study.
* Complete abstinence from sexual intercourse that can result in pregnancy is also acceptable.
* Able to agree to the requirements and restrictions of this study, willing to give voluntary consent, able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

* Female participants who are lactating, pregnant or planning to become pregnant during the study. Carry a diagnosis of diabetes.
* Weigh less than or equal to 80 pounds at any visits.
* Answer "yes" to any of the questions asked on the screening questionnaire (Appendix 10.2.1).
* Have a history of a diagnosis of celiac disease, chronic pancreatitis, steatorrhea, unstable thyroid disease, major affective disorder, psychiatric disorder that required hospitalization in the prior year, immune disorder (i.e., HIV/AIDS), cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit).
* Use any dietary supplements that may impact hydration status within the 30 days prior to the baseline visit (Familiarization Trial/Visit 2).
* Participants must observe a 30-day washout period of no supplementation to be eligible. Consume more than two standard alcoholic drinks per day.
* Use of inhalables, smokables, or the like (e.g., cigarettes, vaporizers, water pipes, or cannabis) within 30 days prior to the first dose of the study product or for the duration of the study.
* Have a medical condition that may impact ability to exercise or ability to ingest prescribed fluid volume. Smoking tobacco products.
* Have a history of alcohol or substance abuse in the 12 months prior to the screening visit.
* Are cognitively impaired and/or unable to give informed consent. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients, or any of the rescue medications.
* Have a current or previous diagnosis with COVID-19 in the three months prior to screening.
* Have had major surgery three months prior to screening or have a planned major surgery during the course of the study.
* Have received or use test product(s) in another research study in the 28 days prior to baseline visit (Familiarization Visit/Visit 2), or longer if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of the current study.
* Have any other active or unstable medical conditions or use medications, supplements, or therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Relative rehydration | Through study completion, an average of 8 weeks
  To determine the effect of the Test Products (TPs) on relative rehydration after exercise, as compared to placebo via percent plasma volume change (hematocrit and hemoglobin) and plasma osmolality

SECONDARY OUTCOMES:
Hydration status | Through study completion, an average of 8 weeks
  To determine the effect of the TPs on hydration status, as compared to placebo via sweat loss
Participant reported outcomes | Through study completion, an average of 8 weeks
  To determine the effect of the TPs on participant reported outcomes, as compared to placebo via bloating, exertion, exhaustion, thermal sensation, feeling of refreshment, stomach upset, and thirst.
Plasma electrolyte levels | Through study completion, an average of 8 weeks
  To determine the effect of the TPs on plasma electrolyte levels, as compared to placebo via sodium, potassium, magnesium, chloride, and calcium.

OTHER OUTCOMES:
Relative effects of dehydration and rehydration | Through study completion, an average of 8 weeks
  To explore the relative effects of dehydration and rehydration from the TPs and control on cognitive function, as compared to placebo via NIH cognitive tool box - Flanker inhibitory control and attention testing performance
Exercise performance | Through study completion, an average of 8 weeks
  To explore the effect of the TPs on exercise performance, as compared to placebo via time to exhaustion

CONTACTS AND LOCATIONS:
Overall Officials: Sean Arent, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No